CLINICAL TRIAL: NCT00990041
Title: Release of Cytokines by Stimulated Peripheral Blood Mononuclear Cells (PBMC) From Chronic Periodontitis Subjects
Status: Completed | Type: Observational
Sponsor: Escola Bahiana de Medicina e Saude Publica (Other)
Collaborators: School of Odontology of Piracicaba - Unicamp (Other)
Other Study IDs: 9002-10-04.PBMC
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Periodontitis
Keywords: periodontitis; find cytokines in blood of periodontal patients
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- PBMC
- periodontitis

SUMMARY:
Background and Objective: It has been reported that peripheral blood mononuclear cells (PBMC) from periodontal patients have a different profile of cytokine release when compared to the ones of healthy patients. Cigarette smoking is a recognized risk factor for periodontitis and is known to affect the systemic and local immune responses. Thus, the aim of the present study was to obtain preliminary data about the interaction of periodontal condition and smoking in the secretion of some cytokines by PBMC.

Material and Methods: PBMC samples were isolated from 19 donors, divided into generalized chronic periodontitis (P; n=10) and periodontal health (H; n=9) groups. In addition, the smokers and non-smokers of each group were separately evaluated: SP- smokers with severe generalized chronic periodontitis (n=5); SH- periodontally healthy smokers (n=5); NSP- non-smokers with severe generalized chronic periodontitis (n=5) and NSH- periodontally healthy non-smokers (n=4). Cells were incubated for 24-48 hours in 500 µL wells containing RPMI 1640 and stimulated with 1.0 ng/mL of E. coli LPS. Supernatants were used to quantify the amounts of TNF-α, IL-6, IL-8 and IL-10 released using ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* periodontitis

Exclusion Criteria:

* diabetes

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy humans
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Odontologia de Piracicaba, Piracicaba, São Paulo, Brazil